CLINICAL TRIAL: NCT00005853
Title: Therapy of Myelodysplastic Syndrome (MDS) With Antithymocyte Globulin (ATG) and TNFR:Fc
Brief Title: Biological Therapy in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1478.00; FHCRC-1478.00; NCI-G00-1793; CDR0000067878 (Registry Identifier: PDQ)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory cytopenia with multilineage dysplasia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Antilymphocyte Serum; Etanercept

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: etanercept

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining different types of biological therapies may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of biological therapy in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of hematologic responses in patients with myelodysplastic syndrome treated with anti-thymocyte globulin and tumor necrosis factor receptor IgG chimera.
* Correlate phenotypic, cytogenetic, and functional disease characteristics with treatment responses in these patients.
* Determine the safety of this treatment regimen in this patient population.

OUTLINE: Patients receive anti-thymocyte globulin IV over 8 hours daily for 4 days followed by tumor necrosis factor receptor IgG chimera subcutaneously twice weekly for 16 weeks.

Patients are followed at 8, 16, and 20 weeks.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndrome with no greater than 20% marrow blasts with:

  * Single or multilineage cytopenia (neutrophils less than 2,000/mm^3 and/or platelet count less than 100,000/mm^3 and/or reticulocyte count less than 18,000/mm^3) OR
  * Transfusion requirement of at least 2 units packed red blood cells per month and one of the following:

    * Suitable marrow donor unavailable
    * Ineligible for a transplantation protocol
    * Unwilling to proceed with transplantation
* No chronic myelomonocytic leukemia

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other severe disease that would preclude study
* No active severe infection (e.g., pneumonia or septicemia) or severe infections within the past 2 weeks

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 4 weeks since prior hematopoietic growth factors
* No concurrent hematopoietic growth factors

Chemotherapy:

* At least 4 weeks since prior cytotoxic therapy
* No concurrent cytotoxic therapy

Endocrine therapy:

* Not specified

Radiation therapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 4 weeks since prior immunomodulatory therapy
* No concurrent immunomodulatory therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-12; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Joachim Deeg, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States